CLINICAL TRIAL: NCT02554890
Title: A Multicenter, Randomized, Double-blind, Double Dummy, Parallel Group, Active-controlled 8-week Study to Evaluate the Effect of Sacubitril/Valsartan (LCZ696) Versus Enalapril on Changes in NT-proBNP and Safety and Tolerability of In-hospital Initiation of LCZ696 Compared to Enalapril in HFrEF Patients Who Have Been Stabilized Following Hospitalization for Acute Decompensated Heart Failure (ADHF).
Brief Title: Comparison of Sacubitril/Valsartan Versus Enalapril on Effect on NT-proBNP in Patients Stabilized From an Acute Heart Failure Episode.
Acronym: PIONEER-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLCZ696BUS01
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-09

CONDITIONS: Acute Heart Failure
Keywords: Acute; Heart Failure; reduced ejection fraction; NTproBNP; Heart failure with reduced ejection fraction (HFREF)
MeSH Terms: conditions — Heart Failure | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sacubitril/valsartan (LCZ696) (Experimental): Initial dose for patients randomized to sacubitril/valsartan (LCZ696) was determined by the blood pressure at the time of randomization. Study treatment was titrated to the target dose of sacubitril/valsartan (LCZ696) 97/103 mg bid (Dose Level 3). Titration was based on blood pressure at the time of the visit. Dose adjustments were only allowed if indicated per protocol defined safety and tolerability criteria and investigator judgement.
  Patients were required to take a total of two tablets twice daily (one tablet of active sacubitril and valsartan and one tablet of enalapril matching placebo pack).
  Interventions: Drug: sacubitril/valsartan (LCZ696); Drug: enalapril matching placebo
- Enalapril (Active Comparator): Initial dose for patients randomized to enalapril were determined by the blood pressure at the time of randomization. Study treatment were titrated to the target dose of enalapril 10 mg bid. Titration were based on blood pressure at the time of the visit. Dose adjustments were only allowed if indicated per protocol defined safety and tolerability criteria and investigator judgement.
  Patients were required to take a total of two tablets twice daily (one tablet of active enalapril, second from sacubitril and valsartan matching placebo pack)
  Interventions: Drug: Enalapril; Drug: sacubitril/valsartan (LCZ696) matching placebo

INTERVENTIONS:
Drug: sacubitril/valsartan (LCZ696) — sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Other Names: LCZ696
  Arms: sacubitril/valsartan (LCZ696)
Drug: Enalapril — Enalapril tablet with minimum dose 2.5 mg, maximum dose 10 mg twice daily administered orally.
  Arms: Enalapril
Drug: sacubitril/valsartan (LCZ696) matching placebo — matching placebo of sacubitril/valsartan (LCZ696) tablet with minimum dose 24/26 mg, maximum dose 97/103 mg twice daily administered orally.
  Arms: Enalapril
Drug: enalapril matching placebo — enalapril matching placebo tablet with minimum dose 2.5 mg, maximum dose 10 mg twice daily administered orally.
  Arms: sacubitril/valsartan (LCZ696)

SUMMARY:
The purpose of this study was to assess the effect of in-hospital initiation of sacubitril/valsartan (LCZ696) vs. enalapril on time averaged proportional change in NT-proBNP in patients who have been stabilized following hospitalization for acute decompensated heart failure (ADHF) and reduced ejection fraction (left ventricular ejection fraction (LVEF) ≤ 40%).

ELIGIBILITY:
Key Inclusion Criteria:

1. Possess the capacity to provide written informed consent which must be obtained before any assessment is performed.
2. Currently hospitalized for ADHF. Patients with a diagnosis of acute heart failure had to have symptoms and signs of fluid overload (i.e. jugular venous distention, edema or rales on auscultation or pulmonary congestion on chest x-ray) at time of hospitalization.
3. Eligible patients will be randomized no earlier than 24 hours and up to ten days after presentation while still hospitalized as long as meet the following definition of stable status:

   * SBP ≥100mm Hg for the preceding 6 hours prior to randomization; no symptomatic hypotension
   * No increase (intensification) in i.v. diuretic dose within last 6 hours prior to randomization
   * No i.v. inotropic drugs for 24 hours prior to randomization
   * No i.v. vasodilators including nitrates within last 6 hours prior to randomization
4. LVEF ≤40% within the past 6 months (including current hospitalization) using echocardiography, multi gated acquisition scan (MUGA), CT scanning, MRI or ventricular angiography, provided no subsequent study documented an EF of >40%.
5. Elevated NT-proBNP ≥ 1600pg/mL OR BNP ≥400 pg/mL during current hospitalization.

Key Exclusion Criteria:

1. Currently taking sacubitril/valsartan tablets or any use within the past 30 days.
2. Enrollment in any other clinical trial involving an investigational agent or investigational device.
3. History of hypersensitivity, known or suspected contraindications, or intolerance to any of the study drugs, including ACEIs, ARBs, or Sacubitril (NEP inhibitor).
4. Patients with a known history of angioedema related to previous ACE inhibitor or ARB therapy.
5. Requirement of treatment with both ACE inhibitor and ARB.
6. eGFR < 30 ml/min/1.73 m2 as measured by the simplified Modification of Diet in Renal Disease (MDRD) formula at screening.
7. Serum potassium > 5.2 mEq/L at screening.
8. Known hepatic impairment (as evidenced by total bilirubin > 3 mg/dL, or increased ammonia levels, if performed), or history of cirrhosis with evidence of portal hypertension such as varices
9. Acute coronary syndrome, stroke, transient ischemic attack; cardiac, carotid or other major CV surgery; percutaneous coronary intervention (PCI) or carotid angioplasty, within one month prior to Visit 1.
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (108):
- United States (108):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fort Smith, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Marino, California
  - Novartis Investigative Site, San Pablo, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Littleton, Colorado
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, West Haven, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Daytona Beach, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lakeland, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Aurora, Illinois
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Oakbrook Terrace, Illinois
  - Novartis Investigative Site, Park Ridge, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Winfield, Illinois
  - Novartis Investigative Site, Elkhart, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Muncie, Indiana
  - Novartis Investigative Site, Richmond, Indiana
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Annapolis, Maryland
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Bay City, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Maplewood, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Camden, New Jersey
  - Novartis Investigative Site, Elmer, New Jersey
  - Novartis Investigative Site, Haddon Heights, New Jersey
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Johnson City, New York
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Poughkeepsie, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Camp Hill, Pennsylvania
  - Novartis Investigative Site, Natrona Heights, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, White River Junction, Vermont
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Lynchburg, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Virginia Beach, Virginia
  - Novartis Investigative Site, Clarksburg, West Virginia
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Ambrosy AP, Duffy CI, McCague K, Hernandez AF, Rocha RA, Braunwald E. Rationale and design of the comParIson Of sacubitril/valsartaN versus Enalapril on Effect on nt-pRo-bnp in patients stabilized from an acute Heart Failure episode (PIONEER-HF) trial. Am Heart J. 2018 Apr;198:145-151. doi: 10.1016/j.ahj.2018.01.004. Epub 2018 Jan 10. PMID 29653636
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Morrow DA, Velazquez EJ, DeVore AD, Desai AS, Duffy CI, Ambrosy AP, Gurmu Y, McCague K, Rocha R, Braunwald E. Clinical Outcomes in Patients With Acute Decompensated Heart Failure Randomly Assigned to Sacubitril/Valsartan or Enalapril in the PIONEER-HF Trial. Circulation. 2019 May 7;139(19):2285-2288. doi: 10.1161/CIRCULATIONAHA.118.039331. No abstract available. PMID 30955360
- [Background] Morrow DA, Velazquez EJ, DeVore AD, Prescott MF, Duffy CI, Gurmu Y, McCague K, Rocha R, Braunwald E. Cardiovascular biomarkers in patients with acute decompensated heart failure randomized to sacubitril-valsartan or enalapril in the PIONEER-HF trial. Eur Heart J. 2019 Oct 21;40(40):3345-3352. doi: 10.1093/eurheartj/ehz240. PMID 31093657
- [Derived] Berardi C, Braunwald E, Morrow DA, Mulder HS, Duffy CI, O'Brien TX, Ambrosy AP, Chakraborty H, Velazquez EJ, DeVore AD; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Black Americans: Data From the PIONEER-HF Trial. JACC Heart Fail. 2020 Oct;8(10):859-866. doi: 10.1016/j.jchf.2020.06.019. Epub 2020 Sep 9. PMID 32919915
- [Derived] Ambrosy AP, Braunwald E, Morrow DA, DeVore AD, McCague K, Meng X, Duffy CI, Rocha R, Velazquez EJ; PIONEER-HF Investigators. Angiotensin Receptor-Neprilysin Inhibition Based on History of Heart Failure and Use of Renin-Angiotensin System Antagonists. J Am Coll Cardiol. 2020 Sep 1;76(9):1034-1048. doi: 10.1016/j.jacc.2020.06.073. PMID 32854838
- [Derived] Berg DD, Braunwald E, DeVore AD, Lala A, Pinney SP, Duffy CI, Gurmu Y, Velazquez EJ, Morrow DA. Efficacy and Safety of Sacubitril/Valsartan by Dose Level Achieved in the PIONEER-HF Trial. JACC Heart Fail. 2020 Oct;8(10):834-843. doi: 10.1016/j.jchf.2020.06.008. Epub 2020 Aug 12. PMID 32800511
- [Derived] DeVore AD, Braunwald E, Morrow DA, Duffy CI, Ambrosy AP, Chakraborty H, McCague K, Rocha R, Velazquez EJ; PIONEER-HF Investigators. Initiation of Angiotensin-Neprilysin Inhibition After Acute Decompensated Heart Failure: Secondary Analysis of the Open-label Extension of the PIONEER-HF Trial. JAMA Cardiol. 2020 Feb 1;5(2):202-207. doi: 10.1001/jamacardio.2019.4665. PMID 31825471
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 964 patients were screened for the study. Of these, 887 patients were randomized, 444 to enalapril and 443 to sacubitril/valsartan, and 875 randomized patients were treated.
Pre-assignment Details: Patients were randomized 1:1 to sacubitril/valsartan or enalapril. At the end of the 8-week treatment period, all patients had a 36-hour washout from study treatment prior to starting the open-label extension to ensure that the blinding of the core study was maintained.
Period: Double-blind
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Started (Randomized) | 444 | 443
Treated Patients (Treated) | 436 | 439
Completed (Continued study treatment during double-blind phase) | 348 | 352
Not Completed | 96 | 91
Not completed — Adverse Event | 45 | 51
Not completed — Death | 6 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Subject/Guardian decision | 21 | 16
Not completed — Lost to Follow-up | 7 | 5
Not completed — Technical problems | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Noncompliance with study treatment | 6 | 5
Period: Open-label
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Started (Randomized) | 0 | 887
Completed (Continued study treatment during open-label phase) | 0 | 835
Not Completed | 0 | 52
Not completed — Adverse Event | 0 | 30
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Subject/Guardian decision | 0 | 11
Not completed — Lost to Follow-up | 0 | 7
Not completed — Technical problems | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are in the Full analysis set (FAS) of treatment groups.
  FAS: Patients who were randomized except those who were not qualified for randomization and have not received study treatment, but were inadvertently randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696) | Total
Number analyzed (Participants) | 441 | 440 | 881
Age, Customized [Number; unit: Participants]
  <65 years | 232 | 253 | 485
  ≥65 years | 209 | 187 | 396
  < 75 years | 363 | 370 | 733
  ≥75 years | 78 | 70 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 113 | 246
  Male | 308 | 327 | 635
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 34 | 75
  Not Hispanic or Latino | 399 | 405 | 804
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Values and Time-averaged Change From Baseline
Description: To assess the effect of in-hospital initiation of sacubitril/valsartan vs. enalapril on the time-averaged percentage change of NT-proBNP from baseline in patients who have been stabilized following hospitalization for ADHF and reduced ejection fraction (left ventricular ejection fraction [LVEF] ≤ 40%) between week 4 and 8.
  Number of patients with both a baseline value and a value at Week 4 or Week 8. Plasma NT-proBNP (pg/mL) values were averaged from Week 4 and Week 8 visits. N-terminal pro b-type natriuretic peptide (NTproBNP) are peptide (small proteins) that are either hormones or part of the peptide that contained the hormone at one time. They are continually produced in small quantities in the heart and released in larger quantities when the heart senses that it needs to work harder, as in heart failure.
Time Frame: Baseline, Week 4 and Week 8
Population: Full analysis set (FAS): consisted of all randomized patients with the exception for those patients who had not been qualified for randomization and had not received study treatment, but had been inadvertently randomized into the study.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
pg/ml | 0.7466 [0.6842 to 0.8147] | 0.5333 [0.4890 to 0.5816]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p < .0001, ANCOVA — ANCOVA model for a log-scaled response with treatment group as a class variable and biomarker baseline value in logarithmic scale as a continuous covariate; expon. back transformed from LS means = 0.7143, 95% CI 2-sided [0.6315 to 0.8080] — Geometric Mean Ratio: Sacubitril/ Valsartan vs. Enalapril

2. Secondary Outcome: Number of Patients With Incidences of Symptomatic Hypotension
Description: Examine the effect of LCZ696 vs. enalapril on incidence of symptomatic hypotension during 8 weeks of treatment Hypotension is low blood pressure. Patients with hypotension may experience symptoms when their blood pressure drops, compared to the patient's normal values. Symptoms of hypotension can include dizziness, lightheadedness, blurred vision, weakness, fatigue, nausea, palpitations, and headache.
Time Frame: 8 weeks of treatment
Population: FAS
Measure: Number; unit: participants
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
participants | 56 | 66

3. Secondary Outcome: Number of Patients With Incidences of Hyperkalemia
Description: Hyperkalemia is defined as Potassium level >5.5 mEq/L. Hyperkalemia is the medical term that describes a potassium level in your blood that's higher than normal. Potassium is a chemical that is critical to the function of nerve and muscle cells, including those in your heart.
Time Frame: 8 weeks of treatment
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Participants | 41 | 51

4. Secondary Outcome: Number of Patients With Incidences of Angioedema
Description: Angioedema is a type of abrupt swelling that occurs under the skin and/or mucous membranes and is often localized to the head, neck, throat, and/or tongue, but may occur elsewhere, including the genitalia and intestines. Severe cases may be associated with difficulty in breathing.
Time Frame: 8 weeks of treatment
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Participants | 11 | 1

5. Secondary Outcome: Change From Baseline in High Sensitivity Troponin (Hs-Troponin)
Description: time-averaged (Weeks 4 and 8) change from baseline in hs-troponin T. hs-Troponin-T is a biomarker that is released from the heart under stress or injury conditions.
Time Frame: Baseline, Week 4/Week 8
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Ratio | 0.7477 [0.6979 to 0.8010] | 0.6345 [0.5920 to 0.6801]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p = 0.0011, ANCOVA; exponentially back transformed from LS m = 0.8487, 95% CI 2-sided [0.7694 to 0.9361] — Geometric Mean Ratio: Sacubitril/ Valsartan vs. Enalapril

6. Secondary Outcome: Change From Baseline in Urinary cGMP
Description: Time-averaged (Weeks 4 and 8) change from baseline in urinary cGMP. Urinary Cyclic GMP (cGMP) is a biomarker measured in the urine that reflects the activity of biomarkers such as BNP (Brain Natriuretic Peptide)
Time Frame: Baseline, Week 4 and Week 8
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Ratio | 0.9641 [0.8832 to 1.0524] | 1.5895 [1.4554 to 1.7359]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p < .0001, ANCOVA; expon. back transformed from LS means = 1.6487, 95% CI 2-sided [1.4559 to 1.8669] — Geometric Mean Ratio: Sacubitril/ Valsartan vs. Enalapril

7. Secondary Outcome: Change From Baseline in Urinary cGMP to Urinary Creatinine Ratio
Description: Time-averaged (Weeks 4 and 8) change from baseline in urinary cGMP to urinary creatinine ratio.
  Urinary cGMP to urinary creatinine ratio is how much urinary cGMP (which reflects natriuretic peptide activity) compared to a compound in the urine called creatinine (which helps your doctor evaluate how well your kidneys are functioning).
Time Frame: Baseline, Week 4 and Week 8
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Ratio | 0.8258 [0.7870 to 0.8665] | 1.1714 [1.1160 to 1.2296]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p < .0001, ANCOVA; expon. back transformed from LS means = 1.4186, 95% CI 2-sided [1.3248 to 1.5190] — Geometric Mean Ratio: Sacubitril/ Valsartan vs. Enalapril

8. Secondary Outcome: Change From Baseline in BNP to NTproBNP Ratio
Description: Time-averaged (Weeks 4 and 8) change from baseline in BNP to NT-proBNP ratio. BNP and NT-proBNP are small proteins produced in large amounts when the heart senses it needs to work harder, such as in heart failure. The test measuring BNP to NT-proBNP is measuring how much of each of these biomarkers are present in order to evaluate heart failure.
Time Frame: baseline, Week 4 and Week 8
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
Ratio | 0.9174 [0.8728 to 0.9642] | 1.3527 [1.2882 to 1.4204]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p < .0001, ANCOVA; expon. back transformed from LS means = 1.4745, 95% CI 2-sided [1.3752 to 1.5810] — Geometric Mean Ratio: Sacubitril/ Valsartan vs. Enalapril

9. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Values and Change From Baseline at Week 8
Description: BNP and NT-proBNP are small proteins produced in large amounts when the heart senses it needs to work harder, such as in heart failure. The test measuring BNP to NT-proBNP is measuring how much of each of these biomarkers are present in order to evaluate heart failure.
  Plasma NT-proBNP (pg/mL) values were Week 8 visit.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Enalapril | Sacubitril/Valsartan (LCZ696)
Number analyzed (Participants) | 441 | 440
pg/ml | 0.6443 [0.5815 to 0.7410] | 0.4596 [0.4150 to 0.5089]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan (LCZ696); Test type: Other; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; expon. back transformed from LS means = 0.7133, 95% CI 2-sided [0.6171 to 0.8245] — Geometric Mean Ratio: Sacubitril/Valsartan vs. Enalapril

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 85 days.
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 85 days.
  Data reported on the safety population.
Groups:
- Double Blind Phase Enalapril: Patients who received Enalapril in the double-blind phase.
- Double Blind Phase Sacubitril/Valsartan: Patients who received Sacubitril/Valsartan in the double-blind phase.
- Open-Label Phase Sacubitril/Valsartan: All patients who received sacubitril/valsartan in the open-label phase.
- Pooled Phase Sacubitril/Valsartan: All patients who received a dose of sacubitril/valsartan either in the double-blind phase or open-label phase.
Arm/Group | Double Blind Phase Enalapril | Double Blind Phase Sacubitril/Valsartan | Open-Label Phase Sacubitril/Valsartan | Pooled Phase Sacubitril/Valsartan
All-Cause Mortality (participants affected / at risk) | 15/436 | 10/439 | 6/828 | 16/851
Serious Adverse Events (participants affected / at risk) | 132/436 | 117/439 | 104/828 | 191/851
Other Adverse Events (participants affected / at risk) | 139/436 | 153/439 | 65/828 | 199/851
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase Enalapril (N=436) | Double Blind Phase Sacubitril/Valsartan (N=439) | Open-Label Phase Sacubitril/Valsartan (N=828) | Pooled Phase Sacubitril/Valsartan (N=851)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 4 | 4 | 2 | 5
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 2 | 4
Angina pectoris (Cardiac disorders) | 3 | 1 | 4 | 5
Angina unstable (Cardiac disorders) | 0 | 2 | 2 | 4
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 5 | 9
Atrial flutter (Cardiac disorders) | 1 | 2 | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 4 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 15 | 7 | 14 | 19
Cardiac failure acute (Cardiac disorders) | 11 | 8 | 10 | 18
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 29 | 16 | 13 | 27
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 3 | 3 | 2 | 5
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 8 | 3 | 3 | 6
Long QT syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 2 | 2
Ventricular tachycardia (Cardiac disorders) | 7 | 5 | 6 | 11
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 2 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Asthenia (General disorders) | 1 | 2 | 2 | 4
Death (General disorders) | 0 | 3 | 2 | 5
Hypothermia (General disorders) | 0 | 1 | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 3 | 3 | 2 | 5
Pain (General disorders) | 0 | 1 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 4 | 1 | 4
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 3 | 2 | 5
Septic shock (Infections and infestations) | 1 | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 1
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 1 | 2
Troponin increased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 10 | 4 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 3
Ketosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 4 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 4 | 5
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 3 | 0 | 3
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 5 | 4 | 9
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 1
Vascular headache (Nervous system disorders) | 1 | 0 | 0 | 0
Lead dislodgement (Product Issues) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 15 | 16 | 5 | 21
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 4 | 1 | 5
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 3 | 2 | 5
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 8 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary ossification (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 2
Extremity necrosis (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypoperfusion (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 17 | 11 | 12 | 21
Orthostatic hypotension (Vascular disorders) | 0 | 3 | 0 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 1
Shock (Vascular disorders) | 0 | 1 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind Phase Enalapril (N=436) | Double Blind Phase Sacubitril/Valsartan (N=439) | Open-Label Phase Sacubitril/Valsartan (N=828) | Pooled Phase Sacubitril/Valsartan (N=851)
Blood creatinine increased (Investigations) | 19 | 30 | 7 | 36
Hyperkalaemia (Metabolism and nutrition disorders) | 39 | 47 | 11 | 57
Dizziness (Nervous system disorders) | 33 | 38 | 17 | 55
Acute kidney injury (Renal and urinary disorders) | 23 | 23 | 3 | 24
Hypotension (Vascular disorders) | 65 | 71 | 33 | 97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02554890/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT02554890/SAP_001.pdf